CLINICAL TRIAL: NCT06557590
Title: Preliminary Study on the Diagnostic Value of 18F-FAPI-04 PET/CT and PET/MR in Patients With Various Types of Malignant Tumors
Brief Title: 18F-FAPI-04 PET/CT and PET/MR in Patients With Various Types of Malignant Tumors
Status: Recruiting | Type: Observational
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Principal Investigator, Hui Ye, Professor, Hunan Cancer Hospital
Other Study IDs: FAPI-002
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Cancer; FAP
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 18F-FAPI-04 — 18F-FAPI-04 was injected into the patients before the PET/CT or PET/MR scans

SUMMARY:
To evaluate the potential usefulness of 18F-FAPI-04 positron emission tomography/computed tomography (PET/CT) and positron emission tomography/magnetic resonance imaging （PET/MR）for the diagnosis of primary and metastatic lesions, detection of recurrence or assessment of pathologic response in various types of cancer.

DETAILED DESCRIPTION:
Subjects with various types of cancer underwent 18F-FAPI-04 PET/CT and PET/MR imaging either for an initial assessment, recurrence detection or assessment of pathologic response. Tumor uptake was quantified by the maximum standard uptake value (SUVmax) and tumor to background (TBR). Using histopathology and follow-up as gold standard, the sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 18F-FAPI-04 PET/CT and PET/MR were calculated.

ELIGIBILITY:
Inclusion Criteria:

patients with suspected or new diagnosed or previously treated malignant tumors (supporting evidence may include MRI, CT, tumor markers and pathology report); patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

patients with non-malignant lesions; patients with pregnancy; the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with suspected or new diagnosed or previously treated malignant tumors.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance | 1 year
  Diagnostic accuracy, The sensitivity, specificity and accuracy of 18F-FAPI-04 PET/CT and PET/MR were calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No